CLINICAL TRIAL: NCT00003096
Title: Molecular Biology of Pediatric Brain Tumors
Brief Title: Gene Testing to Help in the Diagnosis and Treatment of Childhood Brain Tumors
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: B971; COG-B971 (Other: Children's Oncology Group); CCG-B971 (Other: Children's Cancer Group); CDR0000065814 (Other: Clinical Trials.gov)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-08

CONDITIONS: Brain Tumors; Central Nervous System Tumors
Keywords: untreated childhood supratentorial primitive neuroectodermal tumor; untreated childhood medulloblastoma
MeSH Terms: conditions — Brain Neoplasms; Central Nervous System Neoplasms | interventions — Comparative Genomic Hybridization; Cytogenetic Analysis; In Situ Hybridization, Fluorescence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: DNA ploidy analysis
Genetic: comparative genomic hybridization
Genetic: cytogenetic analysis
Genetic: fluorescence in situ hybridization

SUMMARY:
RATIONALE: Analyzing the number and structure of genes found in a child's cancer cells may help doctors improve methods of diagnosing and treating children with brain tumors.

PURPOSE: This clinical trial is studying the number and structure of genes in cancer cells of children with brain tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the chromosomal gains and losses by DNA ploidy analysis and comparative genomic hybridization in patients with primitive neuroectodermal tumors or medulloblastomas.
* Determine the frequency of specific chromosomal abnormalities, including deletions of chromosomal regions 6, 17, and 22, in these patients.
* Perform a statistical analysis to determine possible associations of chromosomal abnormalities and DNA ploidy with patient age, tumor histology, tumor location, extent of disease, and event-free survival.

OUTLINE: DNA ploidy analysis will be performed to determine the overall level of aneuploidy. The results are compared to the comparative genomic hybridization (CGH) analysis, which is used to demonstrate tumor-specific losses or gains, including amplification, of specific chromosomal regions. Tumors are also screened for specific abnormalities by fluorescent in situ hybridization (FISH), which detects chromosomal rearrangements, including balanced translocations, deletions, amplifications, etc. PCR-based microsatellite polymorphism analysis may also be performed.

Primitive neuroectodermal tumors (PNETs) are screened by FISH with a distal 17p13.3 cosmid and a 17q25 cosmid to identify tumors with a 17p deletion. Atypical teratoid/rhabdoid tumors and PNETs without a 17p deletion are screened by FISH with a series of cosmids from 22q11.2. PNETs are also screened by interphase FISH with cosmids from chromosome 6 to identify tumors with deletions.

Patients do not receive the results of the genetic testing and the results do not influence the type or duration of treatment.

PROJECTED ACCRUAL: This study will accrue 360 specimens.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary CNS malignancy consistent with primitive neuroectodermal tumor, medulloblastoma, or atypical teratoid/rhabdoid tumor
* Must be entered on CCG-9921, CCG-9931, CCG-A9961, CCG-99703 or other front-line studies developed from CCG-90024 or CCG-90025
* Retrospective specimens also obtained from CCG-921, CCG-923, CCG-9892, CCG-9921, and CCG-9931

PATIENT CHARACTERISTICS:

Age:

* Under 21

Performance status:

* See Disease Characteristics

Life expectancy:

* See Disease Characteristics

Hematopoietic:

* See Disease Characteristics

Hepatic:

* See Disease Characteristics

Renal:

* See Disease Characteristics

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy

Surgery

* Not specified

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with primitive neuroectodermal tumors / medulloblastoma (PNET/Mb).
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 1996-12; Primary Completion 2006-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Frequency of specific chromosomal gains, losses and rearrangements in a series of infratentorial and supratentorial PNETS
  Estimate the frequency of specific chromosomal gains, losses and rearrangements in a series of infratentorial and supratentorial PNETS diagnosed in children

CONTACTS AND LOCATIONS:
Overall Officials: Jaclyn A. Biegel, PhD, Study Chair — Children's Hospital of Philadelphia
Locations (61):
- United States (56):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Southern California Permanente Medical Group, Downey, California
  - Loma Linda University Cancer Institute at Loma Linda University Medical Center, Loma Linda, California
  - Jonathan Jaques Children's Cancer Center at Miller Children's Hospital, Long Beach, California
  - Samuel Oschin Comprehensive Cancer Institute at Cedars-Sinai Medical Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California
  - Children's Hospital Central California, Madera, California
  - Children's Hospital of Orange County, Orange, California
  - Santa Barbara Cottage Children's Hospital, Santa Barbara, California
  - Children's Hospital Center for Cancer and Blood Disorders, Aurora, Colorado
  - Carole and Ray Neag Comprehensive Cancer Center at the University of Connecticut Health Center, Farmington, Connecticut
  - Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - AFLAC Cancer Center and Blood Disorders Service of Children's Healthcare of Atlanta - Egleston Campus, Atlanta, Georgia
  - Curtis and Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Advocate Lutheran General Cancer Care Center, Park Ridge, Illinois
  - Swedish-American Regional Cancer Center, Rockford, Illinois
  - Simmons Cooper Cancer Institute, Springfield, Illinois
  - St. Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Kosair Children's Hospital, Louisville, Kentucky
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - Breslin Cancer Center at Ingham Regional Medical Center, Lansing, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota
  - Children's Hospitals and Clinics of Minnesota - St. Paul, Saint Paul, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Monmouth Medical Center, Long Branch, New Jersey
  - Carol G. Simon Cancer Center at Morristown Memorial Hospital, Morristown, New Jersey
  - Overlook Hospital, Morristown, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's - Dayton, Dayton, Ohio
  - Tod Children's Hospital, Youngstown, Ohio
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - East Tennessee Children's Hospital, Knoxville, Tennessee
  - Texas Tech University Health Sciences Center School of Medicine - Amarillo, Amarillo, Texas
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
  - Deaconess Medical Center, Spokane, Washington
  - Gundersen Lutheran Center for Cancer and Blood, La Crosse, Wisconsin
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
- Princess Margaret Hospital for Children, Perth, Western Australia, Australia
- Canada (4):
  - Children's & Women's Hospital of British Columbia, Vancouver, British Columbia
  - IWK Health Centre, Halifax, Nova Scotia
  - Allan Blair Cancer Centre at Pasqua Hospital, Regina, Saskatchewan
  - Saskatoon Cancer Centre at the University of Saskatchewan, Saskatoon, Saskatchewan